CLINICAL TRIAL: NCT02278718
Title: A Multicenter, Multinational, Randomized, Controlled, Open Label Study, Performed in Children With Thermal Burns, to Evaluate the Efficacy and Safety of NexoBrid as Compared to Standard of Care (SOC) Treatment
Brief Title: A Study to Evaluate the Efficacy and Safety of NexoBrid in Children With Thermal Burns Compared the Standard of Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MW2012-01-01
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Thermal Burns
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NexoBrid Gel (Experimental): NexoBrid Gel is applied to the burn wound at a dose of 2g or 5g NexoBrid sterile powder mixed with 20g or 50g sterile Gel Vehicle per 180cm^2 of TBSA for four hours.
  Interventions: Drug: NexoBrid
- Standard of Care (Active Comparator): Non surgical and Surgical Debridement
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: NexoBrid — NexoBrid is an enzymatic debriding agent for Eschar Removal.
  Arms: NexoBrid Gel
Procedure: Standard of Care — Surgical or Non-Surgical methods for Eschar Removal
  Arms: Standard of Care

SUMMARY:
This study will be a two-arms study intending to demonstrate superiority of NexoBrid treatment over SOC in children with thermal burns. The study objective is to evaluate the safety and clinical benefit of NexoBrid in hospitalized children (0-17 years) with deep partial and/or full thickness thermal burns of 1-30% TBSA and to compare NexoBrid to standard of care (SOC).

DETAILED DESCRIPTION:
A total of 160 patients will be randomized into NexoBrid and SOC treatment (80 patients per arm).

Age distribution will be managed as follows:

* 45 patients 0-23 months old
* 45 patients 24 months-3 years old
* 30 patients 4-11 years old
* 20 patients 12-17 years old The remaining 20 patients will be enrolled to any of the above groups, per their age during enrollment.

The study will be conducted in three stages. In Stage I, at least 24 children age 4-18 years, hospitalized in burn units, with deep partial thickness burns ranging from 1%-30% TBSA, and who meet the entrance criteria, will be enrolled. Upon completion of stage I, a safety analysis will be performed on safety parameters and the results will be evaluated by a Data Safety Monitoring Board (DSMB) as defined in the agreed charter. If the DSMB does not have any safety concerns, Stage II will commence, this time enrolling at least 26 additional children aged of 1-18 years according to the study procedures. A DSMB will be convened to assess the safety data of the first 50 patients enrolled at stages 1 & 2. If the DSMB has not found any safety concerns, stage III will commence in which patients from the age of birth to 18 years will be included (stage III will include 110 remaining patients required to reach a total of 160 patients).

Following the enrollment of a subject to the study and prior to randomization, physicians will define one or more Target Wounds (TWs) per subject according to TWs definition. All subjects' DPT and FT burns that fit the specified criteria are intended to receive study treatment per randomized study arm and therefore, must be designated as TWs.

Prior to eschar removal treatment with NexoBrid or SOC subjects will be medicated with appropriate analgesia and undergo wound cleansing and dressing of all wounds with antibacterial solutions. Following wound cleansing and antibacterial treatments, subjects will undergo the eschar removal process as per treatment assignment (NexoBrid or SOC, following randomization). Subsequent to eschar removal, all wounds will be assessed and treated in the same manner, in accordance with post-eschar removal wound care strategy. Furthermore, subjects will undergo daily assessments (Vital signs (VS) and pain assessments) for one week and weekly assessments thereafter, until wound closure. Following wound closure, subjects will be followed up at 6 weeks, 12 weeks, and after that, at 6, 12, 18 and 24 months (for a blinded assessment of cosmesis, function and QoL evaluation).

All subjects will be invited to one additional extended follow up visit that will occur at least 30 months after wound closure confirmation for a blinded assessment of cosmesis, function and QoL evaluation.

ELIGIBILITY:
Inclusion Criteria

1. Stage 1: Males and females between 4 years to 18 years of age, Stage 2 (upon DSMB review): Males and females between 1 year to 18 years of age, Stage 3 (upon DSMB review): Males and females between 0 years to 18 years of age.
2. Thermal burns caused by fire/flame, scalds or contact.
3. Patient total burns area ≥ 1% DPT and / or FT,
4. Patient total burns area should be ≤ 30% TBSA; SPT, DPT and/or FT in depth,
5. Signed written informed consent by a legal guardian can be obtained within 84 hours of the burn injury.

At least one wound (a continuous burn area which can be treated in one session; might include several anatomical areas) in a patient should meet all following criteria:

1. Wound that is ≥ 1% TBSA (DPT and/or FT) (not including face, perineal or genital),
2. Wound is composed of DPT and/or FT in depth. Superficial partial thickness areas may be included in the wound area only if cannot be separated from deeper areas (e.g. surrounded by or mixed with DPT areas) and might interfere with the treatment of the deeper areas,
3. Wound that is potentially intended for surgical eschar removal,
4. Wound's blisters can be unroofed, as judged by the investigator.

Exclusion Criteria:

1. Patients weighing less than 3kg,
2. Patients who are unable to follow study procedures and follow up period,
3. Patients with electrical or chemical burns,
4. Patient with a continuous burn area above 15% TBSA,
5. Patients with no DPT and/or FT burn area (only SPT wounds),
6. Patient with circumferential anterior/posterior trunk fire/flame burns, >15% TBSA (Circumferential is defined as encircling ≥ 80% of the trunk circumference),
7. The following pre-enrolment dressings: a. Flammacerium, b. Silver Nitrate (AgNO3),
8. Patients with diagnosed infections,
9. Diagnosis of smoke inhalation injury,
10. Patients with pre-enrolment wounds which are covered by eschar saturated with iodine or by SSD pseudoeschar (e.g. pseudoeschar as a result of >12h SSD treatment),
11. Patients with pre-enrolment escharotomy,
12. Pregnant women (positive pregnancy test) or nursing mothers,
13. Poorly controlled diabetes mellitus (HbA1c>9%),
14. Known Cardio-pulmonary disease, oxygen-dependent pulmonary diseases, broncho-pneumonia, uncontrolled asthma,
15. Known conditions which interfere with circulation (peripheral vascular disease, edema, lymphedema, surgery to the regional lymph nodes, obesity),
16. Any known conditions that would preclude safe participation in the study or adding further risk to the basic acute burn trauma (such as immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder, pulmono-cardiovascular, liver or neoplastic disease),
17. ASA greater than 2
18. Chronic systemic steroid intake,
19. History of allergy and/or known sensitivity to pineapples, papaya, Bromelain or papain,
20. Current (within 12 months prior to screening) suicide attempt,
21. Enrollment in any investigational drug trial within 4 weeks prior to screening,
22. Current (within 12 months prior to screening) alcohol (daily consumption > 3 units for males and >2 units for females) or drug abuse,
23. Prisoners and incarcerated
24. Patients who might depend on the clinical study site or investigator.
25. Patient expresses objection to participate in the study.
26. Patients with other severe cutaneous trauma at the same sites as the burns (i.e. blunt, avulsion or deep abrasion) or previous burn(s) at the same treatment site(s)
27. General condition of patient would contraindicate surgery

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lior Rosenberg, Prof., Study Chair — MediWound Ltd; Yaron Shoham, Dr., Study Director — MediWound Ltd
Locations (36):
- United States (13):
  - Maricopa Special Health Care District, Phoenix, Arizona
  - University Of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - The University of South Florida Board of Trustees, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Shriners Hospital for Children, Boston, Massachusetts
  - Stony Brook University Medical Center, Stony Brook, New York
  - Legacy Emanuel Hospital & Health Center dba Legacy Research Institute, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - Shawn Jekins Children's Hospital, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
- University Hospital, Department of Plastic Surgery, Ghent, Belgium
- S. Khechinashvili University Hospital, Tbilisi, Georgia
- Germany (2):
  - Unfallkrankenhaus Berlin Zentrum für Schwerbrandverletzte mit Plastischer Chirurgie, Berlin
  - Klinikum Stuttgart - Olgahospital, Stuttgart
- Hungary (3):
  - MRE Bethesda Gyermekkórháza, Budapest
  - B.A.Z Megyei Kórház és Egyetemi Oktatókórház, Miskolc
  - Klinikai Kozpont Gyermekgyogyaszati Klinika, Pécs
- India (3):
  - Dr. Ram Manohar Lohia Hospital, Baba Kharak Singh Marg, New Delhi, National Capital Territory of Delhi
  - Krishna Rajendra Hospital, Mysuru
  - Vardhman Mahavir Medical College (VLCC) and Safdarjung Hospital, New Delhi
- Universitary Integrated Hospital Verona (AOUI Verona),, Verona, Italy
- Acute Burn Care &Trauma Surgery, Dept Surgery/Burn Center, Rode Kruis Ziekenhuis, LUMC University Leiden, Beverwijk, Netherlands
- Poland (2):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Szpital Dzieciecy im.prof.dr.med Jana Bogdanowicza, Oddzial Chirurgii i Urologii Dzieciecej z Pododdzialem Leczenia Oparzen, Warsaw
- Romania (2):
  - Spitalul Clinic de Urgenta pentru Copii "Sfanta Maria", Iași
  - Spitalul Clinic de Urgenta Tg- Mures, Târgu Mureş
- Univerzitná nemocnica Bratislava, Klinika popálenin a rekonštrukčnej chirurgie, Bratislava, Slovakia
- Spain (2):
  - La Paz University Hospital, Madrid
  - Boulevar Sur s/n, Valencia
- Ukraine (2):
  - CNPE "City clinical hospital of immediate and urgent medical aid n.a.Meshchaninov" of Kharkiv CC and State institution 'Zaitsev V.T. Institute of general and urgent surgery of the National academy of medical sciences of Ukraine', Kharkiv
  - Communal institution "Odessa Regional Clinical Medical Center", Odesa
- United Kingdom (2):
  - Birmingham Children´s Hospital NHS Foundation Trust, Birmingham
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Background] Rosenberg L, Krieger Y, Bogdanov-Berezovski A, Silberstein E, Shoham Y, Singer AJ. A novel rapid and selective enzymatic debridement agent for burn wound management: a multi-center RCT. Burns. 2014 May;40(3):466-74. doi: 10.1016/j.burns.2013.08.013. Epub 2013 Sep 26. PMID 24074719
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=nexobrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 153 patients that were screened for enrollment, 145 patients were enrolled, randomized and included in FAS analysis. Seven patients were excluded at screening and one patient withdrew consent.
Period: Overall Study
Arm/Group | NexoBrid Gel | Standard of Care
Started | 72 | 73
Treated | 69 | 70
Number of Patients Completed 12 Month FU | 66 | 63
Completed | 66 | 63
Not Completed | 6 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — The patient was randomised but did not receive study drug treatment | 2 | 1
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Overall, 153 patients were screened for enrolment (Enrolled Set). Of the 153 patients enrolled, 145 patients were randomised and included in the FAS: 72 in the NexoBrid treatment arm and 73 in the SOC treatment arm.
Groups:
- Standard of Care (SOC): Non surgical and Surgical Debridement
  Standard of Care: Surgical or Non-Surgical methods for Eschar Removal
- Total: Total of all reporting groups
Arm/Group | NexoBrid Gel | Standard of Care (SOC) | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 5.71 (4.838) | 5.83 (4.909) | 5.77 (4.857)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 42 | 48 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 69 | 66 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 17 | 16 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 51 | 50 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 16.88 (4.368) | 17.09 (4.108) | 16.99 (4.226)

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Eschar Removal (in Days)
Description: Measured by a survival analysis of incidence of complete eschar removal as a function of time.
  Eschar removal will be measured at the end of the debridement starting from randomization date, assessed until complete eschar removal is achieved (in days)
Time Frame: From randomization date until complete eschar removal. For NexoBrid, assessed post application (post 2 h soaking) and for SOC assessed immediately post last dressing change for non-surgical SOC arm and immediately post excision for surgical SOC arm.
Population: All patients who were randomised into the study.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NexoBrid Gel | Standard of Care
Number analyzed (Participants) | 72 | 73
Days | 0.99 [0.88 to 1.4] | 5.99 [2.71 to 9.84]
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care; Wilcoxon test statistic was estimated using generalized Wilcoxon-Gehan test stratified by center group, age group, % TBSA group, proportion of FT area group and number of TWs group. A negative (positive) statistic is associated with longer (shorter) time to the event when treated with NexoBrid vs. Standard of Care. P-value was calculated using the re-randomization test; Test type: Superiority; p = 0.0008, Generalized Wilcoxon-Gehan Test

2. Secondary Outcome: Incidence of Surgical Excision Performed for Eschar Removal
Description: Number of patients who needed surgical excision for eschar removal
Time Frame: Until complete eschar removal has been achieved. Complete eschar removal was achieved within 0.99 days (95% CI: 0.88 to 1.04) for the NexoBrid treatment arm and 5.99 days (95% CI: 2.71 to9.84) for the SOC treatment arm.
Population: Incidence Rate = The proportion and number of patients who required surgical excision for eschar removal.
Measure: Count of Participants; unit: Participants
Arm/Group | NexoBrid Gel | Standard of Care (SOC)
Number analyzed (Participants) | 72 | 73
Participants | 6 | 47
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care (SOC); Incidence of Surgical Excision for Eschar Removal for NexoBrid vs SOC; Test type: Superiority; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 0.025, 95% CI 2-sided [0.007 to 0.090]

3. Secondary Outcome: Blood Loss Related to Eschar Removal
Description: Measured by actual blood loss [ABL]. Actual blood loss was the calculated blood loss summed over all procedures carried out to remove eschar, using hematocrit values measured immediately before each procedure and 4 hours after its completion and the amount of blood transfused was summed over all transfusions carried out during the debridement procedure and up to 24 hours from the end time of the debridement procedure.
Time Frame: Hematocrit - immediately before each procedure and 4 hrs after its completion. The amount of blood transfused will be summed over all transfusions carried out during the debridement procedure and up to 24 hrs from the end time of the debridement procedure
Population: Full analysis set (FAS): 145 patients
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NexoBrid Gel | Standard of Care (SOC)
Number analyzed (Participants) | 72 | 73
mL | 32.26 (284.757) | 202.55 (409.147)
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care (SOC); Test type: Superiority; p = 0.1374, t-test, 2 sided

4. Secondary Outcome: Percent Area of Autograft Performed in DPT Wounds - Main Analysis, Patient Level.
Description: Percent area of deep partial thickness wounds autografted
Time Frame: Assessment will be performed by the investigator immediately after each autograft procedure was performed, before application of coverage.
Population: FAS, Patients with at least one DPT target wound.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | NexoBrid Gel | Standard of Care
Number analyzed (Participants) | 60 | 55
percent | 15.9 (38.57) | 22.8 (43.72)
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care; Test type: Superiority; p = 0.5045, t-test, 2 sided; Mean Difference (Final Values) = -6.9

5. Secondary Outcome: Incidence of Autograft Performed in Deep Partial Thickness Wounds
Description: Number of autografts performed in deep partial thickness wounds
Time Frame: Patient's wounds were assessed until complete healing of all wounds, during the period from complete eschar removal was achieved until complete wound closure. Median time in the population was approx. 4.5 weeks and longest follow up period was of 12 weeks
Population: Main Analysis, Target Wound Level, Deep Partial Thickness Target Wounds Only
Measure: Number; unit: autographs performed
Units Other Than Participants: Deep Partial Thickness Wounds
Arm/Group | NexoBrid Gel | Standard of Care
Number analyzed (Participants) | 72 | 73
Number analyzed (Deep Partial Thickness Wounds) | 81 | 69
autographs performed | 21 | 26
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care; Test type: Superiority; p = 0.0545, t-test, 2 sided; Odds Ratio (OR) = 0.414, 95% CI 2-sided [0.163 to 1.054]

ADVERSE EVENTS:
Time Frame: Time of informed consented until subject's study completion (12 months post wound closure) or earlier if early termination from study.
Description: An adverse event is an undesirable or unintentional event that occurs during use of the study Drug, whether or not considered related to the Drug; this includes clinically significant changes in laboratory values and therapeutic failures. Regardless of the severity or relationship to the investigational Drug, all adverse events occurring during the study period should be recorded in a subject's CRFs.
Arm/Group | NexoBrid Gel | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/69 | 6/70
Other Adverse Events (participants affected / at risk) | 31/69 | 30/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NexoBrid Gel (N=69) | Standard of Care (N=70)
Tachycardia (Cardiac disorders) | 1 | 0
Pyrexia (Gastrointestinal disorders) | 1 | 0
Systemic Inflammatory Response Syndrome (Gastrointestinal disorders) | 1 | 0
Withdrawal Syndrome (General disorders) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Joint Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NexoBrid Gel (N=69) | Standard of Care (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Pain (General disorders) | 4 | 5 — General Disorders and Administration Site Conditions
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 5 | 4
Chills (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3
Ear Infection (Infections and infestations) | 2 | 0
Rhinovirus Infection (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 0 | 2
Haemoglobin Decreased (Investigations) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Bromhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02278718/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT02278718/SAP_001.pdf